CLINICAL TRIAL: NCT07059871
Title: A Prospective, Double-blind, Randomized Controlled Clinical Study of Silkworm Pupa Powder Intervention in the Nutritional Status of Patients With Alzheimer's Disease
Brief Title: A Study of Silkworm Pupa Powder Intervention in the Nutritional Status of Patients With Alzheimer's Disease.
Acronym: AD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZJHIRB-2025-095K
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-05

CONDITIONS: AD - Alzheimer's Disease; Sarcopenia; Asthenia
Keywords: Alzheimer Disease; Sarcopenia; asthenia; nutritional status
MeSH Terms: conditions — Sarcopenia; Asthenia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Silkworm pupa powder, 2 times a day, two packets (12*2 g) each time, take with warm water, before meals, for three months
  Interventions: Dietary Supplement: Silkworm pupa powder
- Control group (Placebo Comparator): Placebo, 2 sachets (12*2 g) twice a day, with warm water, before meals, for three months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Silkworm pupa powder — Silkworm pupa powder, 2 times a day, two packets (12*2 g) each time, take with warm water, before meals, for three months
  Arms: Experimental group
Dietary Supplement: Placebo — Placebo, 2 sachets (12*2 g) twice a day, with warm water, before meals, for three months
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if silkworm pupa powder works to improve the nutritional status of Alzheimer's disease patients. The main questions it aims to answer are:

* Does silkworm pupa powder evaluate the effectiveness of silkworm pupae in improving sarcopenia, frailty and quality of life in AD patients?
* Does silkworm pupa powder improve cognitive function in AD patients?

Researchers will compare silkworm pupa powder to a placebo (a look-alike substance that contains no drug) to see if silkworm pupa powder works to improve the nutritional status of Alzheimer's disease patients.

Participants will:

* Take drug silkworm pupa powder or a placebo every day for 3 months.
* Visit the clinic once every 4 weeks for checkups and tests.
* Keep a diary of their daily consumption.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for probable dementia due to Alzheimer's disease (AD) as defined by the National Institute on Aging and Alzheimer's Association (NIA-AA) (2024).
* Male or postmenopausal female (without childbearing potential). Participants aged 50-90 years (inclusive), with an education level of primary school or higher.
* Mini-Mental State Examination (MMSE) score: ≤17 for illiterate, ≤20 for primary school education, ≤22 for secondary school education, ≤23 for university education; Clinical Dementia Rating (CDR) global score > 2.0.
* Activities of Daily Living (ADL) Scale score >0 and ≤40.
* Nutritional Risk Screening (NRS 2002) score ≥3 at screening/enrollment.
* Good general health status, Eastern Cooperative Oncology Group (ECOG) Performance Status score ≤3.
* If currently receiving approved AD treatments (e.g., acetylcholinesterase inhibitors, GV-971, NMDA receptor antagonists), must be on a stable dose for at least 12 weeks prior to baseline, with stable cognitive assessment scores. Treatment-naïve participants for AD are eligible. Unless otherwise specified, all other permitted concomitant medications (non-AD related) must be stable for at least 4 weeks prior to baseline.
* Availability of a stable, reliable caregiver confirmed by the investigator.
* Voluntarily participate in the clinical study, fully understand and be informed about the study, and sign the Informed Consent Form (ICF); willing and able to comply with and complete all trial procedures. If the participant, in the investigator's judgment, lacks capacity to consent, consent must be obtained according to local laws, regulations, and customs (or signed by the patient's caregiver under the authorization of the patient's legal guardian). Agrees to provide peripheral blood, stool, and urine samples for biomarker analysis during the study.

Exclusion Criteria:

* Dementia caused by: vascular dementia; CNS infections (e.g., AIDS, syphilis); Huntington's disease; Parkinson's disease; Lewy body dementia; traumatic brain injury-related dementia; other physical/chemical factors (e.g., drug intoxication, alcohol intoxication, carbon monoxide poisoning); significant systemic diseases (e.g., hepatic encephalopathy, pulmonary encephalopathy, hypoxic encephalopathy); intracranial space-occupying lesions (e.g., subdural hematoma, brain tumor); endocrine disorders (e.g., thyroid disease, adrenal disease); vitamin deficiencies; or dementia due to any other cause.
* Co-existing autoimmune diseases, such as multiple sclerosis, polymyositis, myasthenia gravis, Guillain-Barré syndrome, ankylosing spondylitis, rheumatoid arthritis, systemic lupus erythematosus, vitiligo, etc.
* Severe renal impairment: Creatinine clearance <30 mL/min (Cockcroft-Gault formula) or other known severe renal disease; Severe hepatic impairment: ALT or AST >10 times the upper limit of normal (ULN), or other known liver diseases such as acute/chronic active hepatitis, cirrhosis, etc.; Acute myocardial infarction or interventional cardiac procedure within 6 months prior to screening; Heart failure (NYHA Class III-IV); Patients with other severe primary neurological, cardiac, pulmonary, hematopoietic, endocrine system diseases, or psychiatric disorders.
* Suspected or confirmed history of alcohol or drug abuse.
* Life expectancy ≤3 months.
* Pregnant or lactating women. Participants of childbearing potential (including male participants engaging in heterosexual intercourse and their female partners of childbearing potential) planning pregnancy or unwilling to use effective contraception from screening initiation until 3 months after discontinuation of the study drug.
* Known allergy/hypersensitivity to any component of the investigational product(s).
* Participation in another investigational drug trial within 30 days prior to screening or current participation in any other clinical trial.
* Presence of any other severe physical or psychiatric illness or laboratory abnormality that may increase the risk associated with study participation or, in the investigator's judgment, makes the patient unsuitable for the study.
* Clinically significant psychiatric disorders or severe psychiatric symptoms.
* MMSE score >26.
* ADL Scale score >40.
* Clinically significant elevation of tumor markers, history of malignancy, or patients with tumors of undetermined nature.
* Significant risk of suicide.
* Chronic alcohol abuse or substance abuse that may interfere with efficacy evaluation.
* Intolerance or allergy to the drugs used in this study.
* Diagnosis of clinically significant cardiovascular or cerebrovascular disease requiring treatment within the past 12 months or current diagnosis.
* Antibiotic use: a. Continuous use of antibiotics for >10 days within 12 weeks prior to baseline; b. Anticipated need for antibiotic treatment exceeding 10 days during the study. Any other disease (e.g., cardiac, respiratory, renal, gastrointestinal diseases potentially affecting absorption such as gastric cancer, gastric bypass surgery, or recurrent diarrhea) not adequately controlled and stable, or any condition the investigator believes may affect participant safety or interfere with study assessments.
* Any other clinically significant abnormality in physical examination, vital signs, laboratory tests, or electrocardiogram (ECG) that, in the investigator's opinion, warrants further investigation or treatment, or may interfere with study procedures or safety.
* Participants with inadequately controlled hemorrhagic disorders (including platelet count <50 x 10^9/L or International Normalized Ratio [INR] >1.5 for participants not on anticoagulant therapy like warfarin).
* Any other condition deemed by the investigator to make the participant unsuitable for study participation.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-23 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | The 4th 、8th and 12th week after taking Silkworm
  Take blood testing and detect hemoglobin levels
Albumin | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Detect blood albumin levels
Serum prealbumin | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Detect serum prealbumin levels
25-hydroxyvitamin D | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Detect blood 25-hydroxyvitamin D levels
Alkaline phosphatase | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Detect blood alkaline phosphatase levels
Parathyroid hormone | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Detect parathyroid hormone levels
Calcitonin | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Detect calcitonin levels
Whole abdominal Computerized tomography (CT) scan | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Take the whole abdominal CT scan
Diagnostic criteria of the 2019 Asian Sarcopenia Working Group | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Evaluate sarcopenia again

SECONDARY OUTCOMES:
Mini-mental State Examination（MMSE） Scale | The 4th、8th and 12th week after taking placebo.
  Take the MMSE Scale again
Clinical Dementia Rating（CDR） Scale | The 4th 、8th and 12th week after taking placebo.
  Take the CDR Scale again
Eastern Cooperative Oncology Group Score | The 4th 、8th and 12th week after taking placebo.
  Take the ECOG Score again
Head Magnetic Resonance Scan | The 4th 、8th and 12th week after taking placebo.
  Take Head MR again
Amyloid β-protein（Aβ） | The 4th 、8th and 12th week after taking placebo.
  Detect the blood Amyloid β-protein levels, include Aβ42、Aβ40、Aβ40/42
Phosphorylated microtubule-associated protein Tau（P-Tau） | The 4th 、8th and 12th week after taking placebo.
  Detect the Phosphorylated microtubule-associated protein Tau levels, include P-tau181、P-tau 217

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Our research is in the exploratory stage and it is not yet clear what results will be obtained.